CLINICAL TRIAL: NCT01245972
Title: A Pilot Study to Examine the Effectiveness of 595nM Pulsed Dye Lasers in the Treatment of Basal Cell Carcinoma and Squamous Cell Carcinoma in Situ
Brief Title: Pilot Study of PDL to Treat BCC and SCCIS
Acronym: PDLNMSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Dr. Shang I. Brian Jiang, Clinical Professor of Dermatology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRPP-101001
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-08

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma in Situ
Keywords: pulsed dye laser; PDL; basal cell carcinoma; squamous cell carcinoma; BCC; SCC; 594nM laser
MeSH Terms: conditions — Carcinoma, Basal Cell; Squamous Intraepithelial Lesions; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): No treatment administered
- PDL Setting 1 (Experimental): PDL Setting 1: 15 J/cm2, 3ms pulse length, no dynamic cooling, 7mm spot size, 10% overlap between the pulses, 2 passes
  Interventions: Procedure: PDL Treatment
- PDL Setting 2 (Experimental): PDL Setting 2: 7.5 J/cm2, 3ms pulse length, no dynamic cooling, 10mm spot size, 10% overlap between the pulses, 2 stacked pulses
  Interventions: Procedure: PDL Treatment

INTERVENTIONS:
Procedure: PDL Treatment — Pulsed-dye laser (PDL) treatment at one of two settings.
  Arms: PDL Setting 1; PDL Setting 2

SUMMARY:
This is a research study to find out more about the use of the pulsed dye laser in the treatment of basal cell carcinoma and early stage squamous cell carcinoma that has not invaded deep into the skin. The purpose of this study is to determine whether the use of the pulsed dye laser (PDL) can completely clear or regress basal cell carcinoma or early stage squamous cell carcinoma.

Pulsed dye laser is a type of laser that is commonly used to treat lesions on the skin that have a prominent blood vessel component. It has been used to treat broken blood vessels on the face, hemangiomas in children and adults, leg veins, port wine stains, and other lesions with a prominent vascular component.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring surgical excision (conventional or Mohs) for biopsy-proven basal cell carcinoma and biopsy-proven squamous cell carcinoma in situ that is clinically present at the pre-operative visit and measures greater than 0.4cm and less than 3cm in size.
* Lesions in the Trunk, Extremities, and Scalp
* Presence of clinically identifiable residual tumor.
* Patients, males and females, aged 18-90 years.
* Willing to participate.
* Able to give informed consent.

Exclusion Criteria:

* Age younger than 18 years
* Location of lesion not in the Trunk, Extremities, and Scalp
* Fitzpatrick skin type V or VI.
* Prior history of known light sensitivity.
* Pregnancy
* Cognitive Impairment
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. I. Brian Jiang, MD, Principal Investigator — UCSD Medical Center, Division of Dermatology

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | PDL Setting 1 | PDL Setting 2
Started | 7 | 8 | 8
Completed | 7 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | PDL Setting 1 | PDL Setting 2 | Total
Number analyzed (Participants) | 7 | 8 | 8 | 23
Age, Continuous [Median (Standard Deviation); unit: years] | 67 (12) | 66 (12) | 56 (12) | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 4 | 4 | 4 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Tumor Clearance
Description: Review of the pathology report showing whether there was residual tumor or not. If there was no residual tumor in the pathology report from the confirmatory excision, the laser treatment was considered successful (tumor clearance).
Time Frame: 21 to 36 days after the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | PDL Setting 1 | PDL Setting 2
Number analyzed (Participants) | 7 | 8 | 8
Participants | 2 | 2 | 5

ADVERSE EVENTS:
Arm/Group | Control | PDL Setting 1 | PDL Setting 2
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 4/8 | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=7) | PDL Setting 1 (N=8) | PDL Setting 2 (N=8)
erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No